CLINICAL TRIAL: NCT06065995
Title: StoMakker: Improving the Quality of Life of Children Receiving an Ileostomy, Colostomy or Continent Urostomy by Offering Access to a Peer Support Platform, Age Dependent Information Provision and Games in a Smartphone Application
Brief Title: StoMakker Mobile Application
Acronym: StoMakker
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: participant inclusion rate could not be achieved timely
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Marlies P. Schijven, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022.0505
Record Dates: First submitted 2023-07-18; First posted 2023-10-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Bowel Diseases; Anorectal Malformations; Spina Bifida; Ostomy
Keywords: Gamification; Mobile application
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anorectal Malformations; Spinal Dysraphism

STUDY DESIGN:
Intervention Model Description: Open-label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to the mobile application
  Interventions: Device: StoMakker
- Control group (No Intervention): Standard care, without access to the application

INTERVENTIONS:
Device: StoMakker — A mobile application that offers age dependent information, a peer support platform and a game
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to investigate if access to the StoMakker application will significantly improve health-related quality of life in children receiving surgery resulting in an ileostomy, colostomy or continent urostomy. The main question it aims to answer are:

* Does access to StoMakker improve health-related quality of life in children receiving surgery for an ostomy?
* Does access to StoMakker improve the anxiety and social functioning of children receiving surgery for an ostomy?
* Does access to StoMakker improve postoperative complications of children receiving surgery for an ostomy?

Participants will be asked to fill in several questionnaires around their surgery. The intervention group of the trial will be given access to the application "StoMakker". The control group of the trial will receive standard care.

DETAILED DESCRIPTION:
Peer support, patient education and -guidance are of crucial importance for children undergoing surgery for a stoma. Current supportive care is either lacking or via paper folders, which is not a suitable strategy for supporting this vulnerable group of children.

The main objective of this prospective trial is to investigate whether access to a peer support platform, age-dependent information provision and games using a smartphone application increases self-reported health related quality of life (HRQOL).

Study population: Children aged between 6 and 18 years old who will receive an ileostomy, colostomy or continent urostomy, are eligible for inclusion. Participants must have access to a smartphone or tablet. Children who are unable to use a smartphone due to mental or physical disabilities will be excluded from the study

Patients and their parents/caregivers are obliged to give written informed consent before they are allowed to be enrolled in the study.

The design of the study is an open-label multicenter randomized controlled trial with a follow-up of 6 months. The intervention group will get access to the app. The control group will receive standard care. Measurement is done via questionnaires, which are send at specificic intervals based on the surgery date. Parents or caregivers will also receive several questionnaires at specific intervals based on the surgery date.

The primary outcome of this study is health-related quality of life. Secondary outcomes are postoperative outcomes, knowledge retention, patient satisfaction with the received care and self-efficacy

ELIGIBILITY:
Inclusion Criteria:

* Individuals scheduled for ileostomy, colostomy or continent urostomy surgery
* Children aged between 6 and 18 years
* Possession of, or continous access to a smartphone or tablet operated with iOS 9 and up or Android 8.0 and up
* Access to email and internet

Exclusion Criteria:

* Incompetence of understanding the Dutch language
* Visual impairment, unless well corrected with visual aids
* Physical disabilities limiting the use of a mobile application
* Mental disabilities limiting the use of a mobile application, learning and filling in questionnaires
* Patients with pre-existing skin conditions such as pemphigus, para-pemphigus or psoriasis that may disturb or influence normal stoma care protocols

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health-related quality of life of participants on the age specific 7 item PROMIS Pediatric Global Health scale (PGH-7) questionnaire at 6 months after surgery | 6 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Global Health scale (PGH-7) is a validated self reported instrument for assessing general health. Scores range from 5 (low health-related quality of life) to 35 (high health-related quality of life). The questionnaire has been translated to dutch and validated in the Netherlands and dutch speaking Belgium
  Change = 6 month score - baseline

SECONDARY OUTCOMES:
Change from baseline in anxiety of participants on the age specific 8 item PROMIS pediatric v2.0 Anxiety and Depressive Symptoms, the short form 8a questionnaire at 6 months follow-up | 6 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) pediatric item banks v2.0 Anxiety and Depressive Symptoms, the short forms 8a is a validated questionnaire. Scores range from 8 to 40 where a higher score indicates a higher level of anxiety
  The questionnaire has been translated to dutch and validated in the Netherlands and dutch speaking Belgium
  Change = 6 month score - baseline
Change from baseline in social functioning of participants on the age specific PROMIS pediatric item bank peer relationships short form 8a at 6 months after surgery | 6 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) pediatric item banks v2.0 Peer relationships, the short forms 8a is a validated questionnaire. Scores range from 8 to 40 where a higher score indicates a higher level of social functioning
  The questionnaire has been translated to dutch and validated in the Netherlands and dutch speaking Belgium
  Change = 6 month score - baseline . Scores range from 8 (low social functioning) to 40 (high social functioning)
Occurrence of any surgery related complications as specified by the clavien-dindo classification within 6 months of follow-up. | 6 months follow up
  The Clavien Dindo Classification is used to rank the severity of a surgical complication. It is based on the type of therapy needed to correct the complication. The scale consists of several grades (Grade I, II, IIIa, IIIb, IVa, IVb and V). Grade I complications are usually mild but Grade II and higher complications are more significant. Examples include (but are not limited to): infections requiring antibiotics, blood transfusions or injury to abdominal or pelvic structures

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No